CLINICAL TRIAL: NCT05925530
Title: A Multicentre, Phase II, Single-Arm, Interventional Study of Neoadjuvant Durvalumab and Platinum-based Chemotherapy (CT), Followed by Either Surgery and Adjuvant Durvalumab or Chemoradiotherapy (CRT) and Consolidation Durvalumab, in Participants With Resectable or Borderline Resectable Stage IIB-IIIB Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study to Assess Neoadjuvant Durvalumab (D) and Platinum-Based Chemotherapy (CT), Followed by Either Surgery and Adjuvant D or CRT and Consolidation D, in Resectable or Borderline Resectable Stage IIB-IIIB NSCLC (MDT-BRIDGE)
Acronym: MDT-BRIDGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9106C00002; 2023-503357-35-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Neoadjuvant; Durvalumab; Chemoradiotherapy; Surgery; Adjuvant; Consolidation; Multidisciplinary team (MDT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Durvalumab will be administered to the participants via intravenous infusion (IV)
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Participants that go on to receive surgery, will receive durvalumab for up to four cycles prior to surgery. Participants that go on to receive CRT will receive durvalumab for up to two cycles prior to CRT. All participants will receive durvalumab every four weeks until disease progression or recurrence or up to 12 months following surgery/CRT, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Other Names: MEDI4736

SUMMARY:
The purpose of this study is to assess efficacy and safety of neoadjuvant durvalumab in combination with platinum-based chemotherapy (CT) given as initial therapy after cancer diagnosis followed by either surgery and adjuvant durvalumab or chemoradiotherapy (CRT) and consolidation durvalumab given alone as further therapy in participants with resectable and borderline resectable stage IIB-IIIB NSCLC.

DETAILED DESCRIPTION:
This will be a multicentre, Phase II, single-arm, global study assessing the efficacy and safety of neoadjuvant durvalumab and platinum-based CT, given intravenously, followed by either surgery and adjuvant durvalumab or definitive CRT and consolidation durvalumab in participants with resectable and borderline resectable stage IIB-IIIB NSCLC.

Neoadjuvant Period A:

All participants will initially receive 2 cycles of neoadjuvant durvalumab + CT (investigator's choice platinum-based) every three weeks. Participants will be assessed for resectability by a multidisciplinary team.

Neoadjuvant Period B:

Cohort 1: Participants who are deemed eligible for surgery will receive study intervention every three weeks for an additional one and up to two cycles, followed by surgery.

CRT:

Cohort 2: Participants with unresectable tumours (according to MDT re-assessment) will receive definitive CRT (6 one-week cycles) for approximately six weeks.

Both cohorts will then go on to receive durvalumab every four weeks until disease progression or recurrence or up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Deemed resectable or borderline resectable at baseline, confirmed by MDT evaluation at diagnosis.
* Previously untreated and pathologically confirmed Stage IIB to select [i.e.N2] Stage IIIB by AJCC v8.
* Nodal status confirmed with whole body FDG-PET and biopsy via endobronchial ultrasound, mediastinoscopy, or thoracoscopy.
* Mandatory brain MRI.
* EGFR and ALK wild-type.
* Medically operable: adequate cardiac and lung function to undergo resection.
* Participant must be ≥ 18 years, at the time of screening.
* Histologically or cytologically documented NSCLC.
* Minimum life expectancy of 12 weeks.
* Minimum body weight of 30 kg.
* Male and female participants must be willing to use acceptable methods of contraception.
* Female participants of childbearing potential must have negative pregnancy test.

Exclusion Criteria:

* Unresectable NSCLC confirmed by MDT evaluation at baseline
* Stage IIIC patients
* Participants whose planned surgery at enrollment is a wedge resection
* Known EGFR mutation or ALK translocation
* Participants contraindicated for surgical intervention due to comorbid conditions
* Participants who are allergic to study intervention.
* Participants with more than one primary tumour.
* Known active hepatitis infection, positive HCV antibody, HBsAg or HBV core antibody (anti-HBc), at screening.
* Female participants who are pregnant or breastfeeding.
* Judgement by the investigator that the participant should not participate in the study.
* Previously infected or tested positive for human immunodeficiency virus.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2027-08-27 (Estimated)

PRIMARY OUTCOMES:
Resection rate | At day of surgery (Within 40 days of the last dose of neoadjuvant treatment)
  Resection rate is defined as the proportion of all participants who underwent definitive surgery. Participants who undergo (ie, start) surgery with the goal of complete tumour resection will be counted as meeting this endpoint.

SECONDARY OUTCOMES:
Resection rate | At the day of surgery (within 40 days after the last dose of neoadjuvant treatment)
  Resection rate will be further assessed separately in participants deemed resectable at baseline and participants deemed borderline resectable at baseline.
R0, R1, R2 resection rates | At the day of surgery (within 40 days after the last dose of neoadjuvant treatment)
  The R0, R1, and R2 resection rates (assessed separately) are defined as the proportion of resected participants with resection margins assessed as R0, R1, and R2 respectively. R0 corresponds to resection for cure or complete remission, R1 to microscopic residual tumour, R2 to macroscopic residual tumour.
Pathological complete response (pCR) | At the day of surgery (within 40 days after the last dose of neoadjuvant treatment)
  pCR will be defined as the proportion of participants who undergo surgery and have 0% residual viable tumour cells in resected lung and lymph nodes.
Overall Survival (OS) | From first dose of study intervention until death, withdrawal of consent, or the end of the study (approximately 3.5 years)
  OS will be defined as the time from first dose of study intervention until the date of death due to any cause.
Overall Survival (OS) rate | At 12 months and 24 months
  The proportion of participants alive at 12 and 24 months.
Event-free survival (EFS) | From first dose of study intervention until progression of disease (PD), recurrence or death, withdrawal of consent, or the end of the study (approximately 3.5 years)
  EFS is defined as the time from the first dose of study intervention to any of the following events: PD that precludes surgery, progression or recurrence of disease after surgery, PD in the absence of surgery, disease progression, recurrence, or death due to any cause.
Event-free survival (EFS) rate | At 12 months and 24 months
  The proportion of participants alive and event-free at 12 and 24 months.
Progression Free Survival (PFS) | From first dose of study intervention until disease progression, death, withdrawal of consent, or the end of the study (approximately 3.5 years)
  PFS is defined as the time from the first dose of study intervention to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.-defined PD, as assessed by the investigator, or death due to any cause.
Progression Free Survival (PFS) rate | At 12 months and 24 months
  The proportion of participants alive without disease progression at 12 and 24 months.
Objective response rate (ORR) pre-surgery/pre-chemoradiotherapy (CRT) | From first dose of study intervention until death, surgery/start of CRT
  ORR is defined as the proportion of participants who have unconfirmed complete response or partial response as assessed by the investigator per RECIST 1.1.
ORR during study intervention and definitive CRT | From MDT re-assessment timepoint (baseline for this endpoint) until the first tumour assessment after definitive CRT
  ORR is defined as the proportion of participants who have unconfirmed complete response or partial response as assessed by the investigator per RECIST 1.1.
Percentage of all participants with circulating tumor DNA (ctDNA) clearance | From Cycle 1 Day 1 up to pre-surgery/CRT (within 7 to 14 days pre-surgery/CRT) [Each cycle is of 3 weeks]
  Circulating tumour DNA clearance (ie, cMR) will be defined as a change from detectable ctDNA to undetectable ctDNA (ctDNA concentration less than limit of detection) at specified timepoints. The percentage of all biomarker-evaluable participants with ctDNA clearance will be assessed.
Number of participants with adverse events | From enrollment up to at least 90 days after last dose of study intervention
  Safety and tolerability will be evaluated in terms of adverse events and serious adverse events.
Surgical safety: Duration of surgical procedure | Time from start of surgery to end of surgery
  The safety of study intervention will be evaluated from start to end of surgery
Surgical safety: Length of post operative hospital stay | Time from the beginning of the surgery/procedure to the discharge of hospital
  The safety of study intervention will be evaluated during post operative hospital stay
Surgical safety: Intended surgical approach | At baseline
  Intended surgical approach at baseline (minimally invasive vs open thoracotomy).
Surgical safety: Actual surgical approach | At surgery
  Actual surgical approach (minimally invasive vs open thoracotomy).
Surgical safety: Intended surgical procedure | At baseline
  Intended surgical procedure (lobectomy vs bilobectomy vs sleeve resection vs pneumonectomy).
Surgical safety: Actual surgical procedure | At surgery
  Actual surgical procedure (lobectomy vs bilobectomy vs sleeve resection vs pneumonectomy)
Number of participants with delayed surgery | 40 days after last dose of study intervention to surgery
  The safety of study intervention will be evaluated for participants with delayed surgery
Surgical safety: Length of surgical delays | 40 days after last dose of study intervention to surgery
  The safety of study intervention will be evaluated during the length of the surgical delay
Number of participants with reason of surgical delay | 40 days after last dose of study intervention to surgery
  The safety of study intervention will be evaluated for participants with reason of surgical delay
Time from last neoadjuvant dose to surgery | Time from last neoadjuvant dose of study intervention to surgery
  The safety of the study intervention will be evaluated from last neoadjuvant dose to surgery

CONTACTS AND LOCATIONS:
Locations (42):
- United States (3):
  - Research Site, The Bronx, New York
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
- Research Site, Vienna, Austria
- Canada (3):
  - Research Site, Kingston, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- France (8):
  - Research Site, La Tronche
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Mulhouse
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Großhansdorf
  - Research Site, Moers
  - Research Site, Würzburg
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Törökbálint
- Italy (7):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Peschiera del Garda
- Research Site, Lisbon, Portugal
- Spain (7):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (2):
  - Research Site, Solna
  - Research Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies-sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/